CLINICAL TRIAL: NCT00967499
Title: A Multi-Center, Open-Label, 2-Arm, Randomized, Stratified, Parallel, Pilot Study to Assess Palonosetron vs. Ondansetron as Rescue Medication in Subjects That Develop Postoperative Nausea and Vomiting (PONV) in the Postanesthesia Care Unit (PACU)
Brief Title: Pilot Study to Assess Palonosetron Versus Ondansetron as Rescue Medication in Subjects That Develop Postoperative Nausea and Vomiting (PONV) in the Postanesthesia Care Unit (PACU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALO-08-11
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; rescue
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ondansetron
- 2 (Active Comparator)
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Ondansetron — Subjects will receive ondansetron 4 mg intravenously (IV) and will be followed for 72 hours.
  Ondansetron is a selective 5-HT3 receptor antagonist. It is indicated for the prevention of nausea and vomiting associated with initial and repeat courses of emetogenic cancer chemotherapy, including high-dose cisplatin and prevention of postoperative nausea and/or vomiting.
  Other Names: Zofran
  Arms: 1
Drug: Palonosetron — Subjects will receive palonosetron HCl 0.075 mg IV and will be followed for 72 hours.
  Palonosetron hydrochloride (Aloxi®) is a potent and selective 5-HT3 receptor antagonist for the prevention of acute nausea and vomiting associated with initial and repeat courses of moderately and highly emetogenic cancer chemotherapy, the prevention of delayed nausea and vomiting associated with initial and repeat courses of moderately emetogenic cancer chemotherapy, and the prevention of postoperative nausea and vomiting for up to 24 hours following surgery.
  Other Names: Aloxi
  Arms: 2

SUMMARY:
The purpose of this study is to investigate palonosetron versus ondansetron as rescue medication in subjects that develop postoperative nausea and vomiting (PONV) in the Postanaesthesia Care Unit (PACU).

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a frequent complication of surgery, which can lead to subject discomfort and dissatisfaction as well as considerable subsequent medical and economic consequences. In this multi-center, open-label, parallel, randomized, pilot study, outpatient surgical patients who experience post-operative nausea or vomiting in the PACU will be stratified by gender and randomly assigned to either palonosetron HCl 0.075 mg IV or ondansetron 4 mg IV in a minimization random allocation. Male or female outpatients, scheduled for elective laparoscopic abdominal or gynecological surgery under general endotracheal anesthesia will be enrolled. All subjects will be asked to attend 2 visits to the study center:

1. Screening (Days -14 to -1)
2. Treatment (Day 1, the day of the surgical procedure and randomization) Subjects treated will receive a follow-up telephone call by the Study Coordinator on Study Day 4 or 5 to review the subject diary for completion, to review adverse events, and concomitant medications, prior to the subject returning the completed diary to the site.

At the Screening visit, subjects who provide their informed consent will undergo a clinical assessment. Demographic and baseline characteristics, including entrance criteria determination, medical history, history of PONV and/or currently prone to motion sickness, smoking status, prior and concomitant medication, physical examination, and vital signs will be documented.

On the day of surgery, all subjects who meet the eligibility criteria will be prophylactically treated prior to anesthesia with ondansetron 4 mg IV, as preoperative antiemetic treatment. As clinically indicated for rescue therapy, subjects experiencing a nausea severity score ≥4 on the 11-point NRS, vomiting, or indicating a subject request will receive blinded study medication as their first line rescue therapy for PONV while in the PACU and no more than 6 hours after PACU admission. Subjects requiring rescue medication need to be dosed within 10 minutes of identifying the need for rescue medication. In an effort to ensure that this timeline is not exceeded, the sites will be allowed to randomize the subject prior to surgery, on the day of surgery. Subjects who are randomized but do not require rescue therapy and therefore not dosed with study drug, will be considered 'Subjects randomized but not treated'.

Subject diaries will be used to record the date and time of study drug administration, the reason for administering rescue medication, baseline emetic symptoms immediately prior to administration of rescue medication, the occurrence of emetic episodes, the severity and duration of nausea, and subject functioning evaluations for nausea and emesis assessed according to the modified Osoba questionnaire (Martin et. al. 2003). The baseline assessment that is performed just prior to administering the rescue medication must indicate that at least one of the following conditions was met:

1. the subject had a nausea severity score ≥4 on the 11-point (0-10) NRS
2. vomiting
3. subject request: subject request must be approved by site staff and must be based on either nausea or emesis symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >=18 years of age.
2. American Society of Anesthesiologists (ASA) physical status 1 to 3.
3. Presence of at least 2 of the following PONV risk factors:

   * female gender
   * history of PONV and/or currently prone to motion sickness (if the subjects cannot remember their last experience of motion sickness or if they suffered from it as a child, then they will not be classified as "prone")
   * non-smoking status (never smoked or quit >=12 months ago)
4. Outpatient undergoing elective laparoscopic gynecological or abdominal surgery
5. Surgery for which anesthesia is expected to last at least 30 minutes
6. General endotracheal anesthesia conducted as outlined in the anesthetic procedures section of the protocol
7. If a subject has a known hepatic, renal or cardiovascular impairment, he/she may be enrolled in this study at the discretion of the Investigator
8. If a subject has or may develop prolongation of cardiac conduction intervals, particularly QTc, he/she may be enrolled at the discretion of the Investigator.
9. If a subject is female of childbearing potential, she must be using reliable contraceptive measures and have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test within 72 hours prior to surgery on Day 1. Reliable contraceptive measures include implants, injectables, combined oral contraceptives, some intrauterine devices, vasectomized partner or sexual abstinence. Non-childbearing potential is defined as post-menopausal for at least 2 years or documented surgical sterilization or hysterectomy at least 3 months before study start.

Exclusion Criteria:

1. Inability to understand or cooperate with the study procedures as determined by the Investigator.
2. Women who are pregnant, nursing or planning to become pregnant, are not using effective birth control, or that have had a positive serum pregnancy test within 72 hours prior to surgery on Day 1.
3. A cancer patient who has had chemotherapy within 4 weeks prior to study entry (Screening visit).
4. Any kind of emetogenic radiotherapy within 8 weeks prior to study entry (Screening visit).
5. Has received any investigational drugs within 30 days before study entry.
6. Having taken any drug with potential antiemetic efficacy within 24 hours prior to anesthetic procedures.
7. Any vomiting, retching, or nausea in the 24 hours preceding the administration of anesthesia .
8. Body mass index (BMI) > 40.
9. Known or suspected current history of alcohol abuse or drug abuse.
10. Known hypersensitivity/contraindication to 5-HT3 antagonists or study drug excipients.
11. Epileptic patients.
12. Any condition, which in the opinion of the Investigator would make the subject ineligible for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2009-07-13 (Actual); Primary Completion 2009-12-18 (Actual); Study Completion 2009-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Precision Trials, Phoenix, Arizona
  - Accurate Clinical Trials, Inc, Laguna Hills, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Derived] Candiotti KA, Ahmed SR, Cox D, Gan TJ. Palonosetron versus ondansetron as rescue medication for postoperative nausea and vomiting: a randomized, multicenter, open-label study. BMC Pharmacol Toxicol. 2014 Aug 16;15:45. doi: 10.1186/2050-6511-15-45. PMID 25127659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States from 13 July 2009 to 18 December 2009. PONV is postoperative nausea and vomiting and PACU is postanesthesia care unit.
Pre-assignment Details: A total of 239 participants were enrolled and screened, of which 19 participants were screen failures and 220 participants were randomized out of which only 98 participants received the treatment. 122 randomized participants were not treated as they did not experience PONV within 6 hours of PACU admission.
Groups:
- Palonosetron: Participants received a single dose of palonosetron 0.075 milligram (mg), intravenously, over a period of 10 seconds as preoperative antiemetic treatment prior to anesthesia administration on Day 1 (day of surgical procedure). Participants had also received same treatment as rescue medication up to 72 hours post-surgical procedure if experienced PONV.
- Ondansetron: Participants received a single dose of ondansetron 4 mg, intravenously, over a period of 30 seconds as preoperative antiemetic treatment prior to anesthesia administration on Day 1 (day of surgical procedure). Participants had also received same treatment as rescue medication up to 72 hours post-surgical procedure if experienced PONV.
Period: Overall Study
Arm/Group | Palonosetron | Ondansetron
Started | 111 | 109
Treated (Full Analysis Set) | 48 | 50
Completed | 46 | 49
Not Completed | 65 | 60
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Sponsor Decision | 1 | 0
Not completed — Randomized but not treated | 63 | 59

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were randomly assigned to and received study medication.
Groups:
- Palonosetron: Participants received a single dose of palonosetron 0.075 mg, intravenously, over a period of 10 seconds as preoperative antiemetic treatment prior to anesthesia administration on Day 1 (day of surgical procedure). Participants had also received same treatment as rescue medication up to 72 hours post-surgical procedure if experienced PONV.
- Total: Total of all reporting groups
Arm/Group | Palonosetron | Ondansetron | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.22) | 42.5 (13.80) | 41.8 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 38 | 45 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 36 | 36 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Control
Description: Complete control was defined as participants with no emetic episode, no rescue medication, and no more than 3 on the nausea numeric rating scale (NRS) severity score. The 11-point NRS scale (ranging from 0-10), where 0 means no nausea, 2 or 3 was mild nausea, around 5 was moderate nausea, 7 and higher was severe nausea and 10 means the worst possible nausea. Higher scores were considered as worse outcome.
Time Frame: Up to 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 48 | 50
percentage of participants | 25.0 | 18.0
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; Test type: Superiority; p = 0.4010, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With Complete Response
Description: Complete response was defined as participants with no emetic episode and no use of rescue medication. An emetic episodic is defined as any number of retches (unproductive emesis) in a single 5-minute period; 1 or a sequence of vomits in a close succession not relieved by a period of relaxation of at least 2 minutes; or retching of less than (<) 5 minutes duration combined with a single vomit.
Time Frame: Up to 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 48 | 50
percentage of participants | 31.3 | 26.0
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; Test type: Superiority; p = 0.5672, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants Who Did Not Experience Any Episode of Emesis
Time Frame: Up to 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 48 | 50
percentage of participants | 70.8 | 52.0
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; Test type: Superiority; p = 0.0570, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants Who Did Not Receive Any Rescue Medication Post-surgical Procedure
Time Frame: Up to 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 48 | 50
percentage of participants | 37.5 | 44.0
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; Test type: Superiority; p = 0.5150, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Nausea Severity Score
Description: Severity of nausea was assessed at specific time points using an 11-point NRS scale (ranging from 0-10) for evaluation of nausea severity. On the 0-10 rating scale, 0 means no nausea, 2 or 3 was mild nausea, around 5 was moderate nausea, 7 and higher was severe nausea and 10 means the worst possible nausea. Higher scores were considered as worse outcome.
Time Frame: Baseline up to 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication. Here overall number of participants analyzed "N" signifies participants who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 47 | 48
score on a scale
  Baseline | 5.7 (1.84) | 5.9 (1.86)
  Change at 72 hours postdose: number analyzed (Participants) | 47 | 46
  Change at 72 hours postdose | -5.1 (2.36) | -5.6 (2.25)
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; Test type: Superiority; p = 0.3601, Cochran-Mantel-Haenszel — P-values are based on Cochran-Mantel-Haenszel row mean score test with gender adjustment for the ranks of the change from baseline values

6. Secondary Outcome: Modified Osoba Nausea and Emesis Module Questionnaire Score
Description: Modified Osoba nausea and emesis module questionnaire was used to assess the impact of nausea and emesis on functional interference at 24, 48 and 72 hours postdose. The modified Osoba questionnaire included specific questions regarding the interference of nausea and emesis in daily activities (appetite, sleep, physical activities, social life, and enjoyment of life) with respective choices. The raw score of the modified Osoba questionnaire was the arithmetic mean of the non-missing item scores, using 1 for the answer "not at all", 2 for the answer "a little", 3 for the answer "quite a bit", and 4 for the answer "very much". Raw score range from 5-20 and the total score was computed by linearly transformed the raw score to final score range as 0 to 100 by calculating ([RS-1]/range)*100, with RS being the raw score and range being 3 in this case of answers scored from 1 to 4. Lower scores indicate better quality of life.
Time Frame: 24, 48 and 72 hours postdose
Population: The full analysis set included all participants who were randomly assigned to and received study medication. Here "overall number of participants analyzed" are participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Palonosetron | Ondansetron
Number analyzed (Participants) | 47 | 47
score on a scale
  24 Hours Postdose | 11.3 (27.38) | 12.1 (23.94)
  48 Hours Postdose | 6.5 (19.29) | 7.0 (18.44)
  72 Hours Postdose | 6.7 (17.80) | 6.2 (15.25)
Statistical Analysis 1: Comparison: Palonosetron vs Ondansetron; 24 hours postdose; Test type: Superiority; p = 0.3453, Mann-Whitney Test
Statistical Analysis 2: Comparison: Palonosetron vs Ondansetron; 48 hours postdose; Test type: Superiority; p = 0.7874, Mann-Whitney Test
Statistical Analysis 3: Comparison: Palonosetron vs Ondansetron; 72 Hours Postdose; Test type: Superiority; p = 0.8485, Mann-Whitney Test

ADVERSE EVENTS:
Time Frame: From on or after date of first dose of study drug up to and including 30 days after last dose of study drug, or up to approximately 158 days
Arm/Group | Palonosetron | Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 6/48 | 8/50
Other Adverse Events (participants affected / at risk) | 43/48 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=48) | Ondansetron (N=50)
Extrasystoles (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Pain management (Surgical and medical procedures) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=48) | Ondansetron (N=50)
Bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Eye swelling (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Uvulitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Chills (General disorders) | 1 | 2
Irritability (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Pnuemonia (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 37 | 42
Incision site oedema (Injury, poisoning and procedural complications) | 1 | 0
incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 3 | 4
Dizziness postural (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes